CLINICAL TRIAL: NCT07362303
Title: Neuralert Stroke Monitor Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neuralert Technologies LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 859883
Record Dates: First submitted 2025-12-08; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Surgery; Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cardiac Surgery Patients (Experimental): Device: Neuralert Monitor Device to identify upper extremity asymmetry in patients who are high risk for stroke.
  Interventions: Device: Neuralert Monitor

INTERVENTIONS:
Device: Neuralert Monitor — The Neuralert monitoring system, a non-invasive device worn on each wrist, is designed to provide continuous monitoring for asymmetry in the extremities, sending an alert to healthcare workers upon identification, thus expediting recognition of stroke.

SUMMARY:
The Neuralert monitoring system, a non-invasive device worn on each wrist, is designed to provide continuous monitoring and expedited recognition of stroke by identifying asymmetry in the extremities, facilitating patient treatment and improving outcomes. This study is designed to evaluate the safety and effectiveness of the Neuralert Monitor. This study aims to show that the device produces fewer than 2 false alarms per patient per day on average, and that the device detects stroke with a sensitivity significantly greater than a device producing 2 random alerts per day.

ELIGIBILITY:
Inclusion Criteria: (all must be yes)

1. Male or female age ≥ 22 years
2. Admitted or planned admission to one of the participating hospitals and followed by the Cardiothoracic (CT) Surgery or Vascular Surgery services
3. Considered at high risk for stroke while in the hospital based on:

   * Interventions or procedures that are high-risk for stroke performed during the hospitalization, which may include:

     * Intracardiac surgical or endovascular procedures, including valve replacement
     * Ascending aorta or aortic arch surgical or endovascular repair
     * Open surgical or endovascular carotid revascularization
   * Other cardiac procedures along with a high-risk medical history:

     * Age ≥ 80 years
     * Prior stroke/ transient ischemic attack (TIA)
     * Hypercoagulable state (i.e., prior clotting events attributed to active malignancy or a diagnosed thrombophilia) requiring lifelong anticoagulation
     * Severely reduced left ventricular cardiac ejection fraction (i.e., <30%) or anterior left ventricular wall akinesis
     * Atrial fibrillation

Exclusion Criteria: (all must be no)

1. Any medical or psychological conditions that, in the opinion of the investigator, would compromise the subject's safety or successful participation in the study
2. Baseline preoperative asymmetric upper extremity weakness as assessed by the Investigator, defined as a differential in the NIHSS upper extremity motor score between the two arms of >0
3. Above the wrist amputation
4. Unwilling to provide informed consent or no legally authorized representative willing to provide consent if the patient is unable
5. Currently imprisoned

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2028-01-15 (Estimated); Study Completion 2028-07-15 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Device | through study completion, an average of 2 years
  To show that the sensitivity of the Neuralert Monitor exceeds the specified performance goal, and
Safety of Device | through study completion, an average of 2 years
  To show that the mean number of false alarms/patient/day for the Neuralert Monitor is less than the specified performance goal.

SECONDARY OUTCOMES:
Length of time to detection of any stroke | through study completion, an average of 2 years
  Time from last known normal to detection of any stroke with weakness
Length of time to detection of stroke by Neuralert | through study completion, an average of 2 years
  Time from last known normal to detection by the Neuralert Monitor of any stroke with weakness
Number of alerts caused by stroke (PPV) | through study completion, an average of 2 years
  How often an alert is caused by confirmed stroke

OTHER OUTCOMES:
Number and type of causes of false alarms | through study completion, an average of 2 years
  A false alarm is defined as any alarm that does not result in a clinical diagnosis of stroke after the next evaluation by the clinical team
Sensitivity of device | through study completion, an average of 2 years
  Sensitivity of device for detection of any stroke, regardless of whether the stroke includes asymmetric weakness
Number of care visits | through study completion, an average of 2 years
  Number of usual care visits documented in the electronic health record
Number and type of adverse events | through study completion, an average of 2 years
  Any adverse events collected during the study

REFERENCES:
- [Background] Messe SR, Kasner SE, Cucchiara BL, McGarvey ML, Cummings S, Acker MA, Desai N, Atluri P, Wang GJ, Jackson BM, Weimer J. Derivation and Validation of an Algorithm to Detect Stroke Using Arm Accelerometry Data. J Am Heart Assoc. 2023 Feb 7;12(3):e028819. doi: 10.1161/JAHA.122.028819. Epub 2023 Jan 31. PMID 36718858